CLINICAL TRIAL: NCT07148622
Title: Randomized Controlled Trial on the Effects of Different Antibiotic Regimens in Preterm Premature Rupture of Membranes After 34 Weeks
Brief Title: Effects of Different Antibiotic Regimens in Preterm Premature Rupture of Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Onur Karaaslan, YuzuncuYıl, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VYYU-KHD-OK-11
Record Dates: First submitted 2025-08-16; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Preterm Premature Rupture of Membranes (PPROM); Prophylaxis; Perinatal Outcomes
Keywords: Preterm premature rupture of membranes, prophylaxis, perinatal outcomes
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes | interventions — Ampicillin; Azithromycin; Clarithromycin; Amoxicillin

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotic regimen 1 (Active Comparator)
  Interventions: Drug: Antibiotic regimen 1: sulbactam + ampicillin + azithromycin
- Antibiotic regimen 2 (Active Comparator)
  Interventions: Drug: Antibiotic regimen 2: ceftriaxone + clarithromycin + amoxicillin

INTERVENTIONS:
Drug: Antibiotic regimen 1: sulbactam + ampicillin + azithromycin — For the first 48 hours, 4×2 g IV sulbactam + ampicillin, 1 g oral azithromycin on day 1, and from days 3-7, 3×500 mg oral amoxicillin
  Arms: Antibiotic regimen 1
Drug: Antibiotic regimen 2: ceftriaxone + clarithromycin + amoxicillin — For the first 48 hours, 1×1 g IV ceftriaxone + 2×500 mg oral clarithromycin, and from day 3 onwards, 3×500 mg oral amoxicillin + 2×500 mg oral clarithromycin.
  Arms: Antibiotic regimen 2

SUMMARY:
To investigate the effects of different antibiotic regimens used in preterm premature rupture of membranes (PPROM) on maternal and fetal outcomes after 34 weeks of gestation.

DETAILED DESCRIPTION:
Background: To investigate the effects of different antibiotic regimens used in preterm premature rupture of membranes (PPROM) on maternal and fetal outcomes after 34 weeks of gestation.

Methods: A total of 40 pregnant women diagnosed with PPROM after the 34th week of gestation were included in the study and randomly divided into two equal groups. Group-1: Sulbactam + ampicillin, azithromycin, and amoxicillin. Group-2: Ceftriaxone, clarithromycin, and amoxicillin. For all cases, obstetric history, time of delivery, latency period, infection markers, neonatal birth weight, APGAR scores, NICU requirement and length of stay, type of delivery and maternal complications were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies,
* PPROM after 34 weeks of gestation

Exclusion Criteria:

* Patients with fetal anomalies
* Preeclampsia, gestational or pregestational diabetes mellitus,
* Multiple pregnancies,
* Chorioamnionitis, placental abruption, cord prolapse, fetal distress, or other complicated pregnancies.
* Maternal immunodeficiency
* The presence of other infections requiring antibiotic therapy, antenatal corticosteroid use, chronic diseases,
* Unwillingness to participate and sign the detailed informed consent form

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-10 (Actual)

PRIMARY OUTCOMES:
mode of birth checklist | From enrollment to the end of treatment at 4 weeks"
  Effect of different antibiotic regimens on fetal and maternal outcomes: mode of birth checklist
neonatal birth weight | From enrollment to the end of treatment at 4 weeks"
  neonatal birth weight
1st and 5th minute APGAR scores | From enrollment to the end of treatment at 4 weeks"
  1st and 5th minute APGAR scores
need for NICU (neonatal intensive care unit) admission | From enrollment to the end of treatment at 4 weeks"
  need for NICU (neonatal intensive care unit) admission
duration of NICU stay | From enrollment to the end of treatment at 4 weeks"
  duration of NICU stay.
White blood cell (WBC) count | From enrollment to the end of treatment at 4 weeks"
  White blood cell (WBC) count was measured every 48 hours
C-reactive protein (CRP) levels | From enrollment to the end of treatment at 4 weeks"
  C-reactive protein (CRP) level was measured every 48 hours
Maternal complications | From enrollment to the end of treatment at 4 weeks"
  Maternal complications; chorioamnionitis, placental abruption

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Lee J, Romero R, Kim SM, Chaemsaithong P, Yoon BH. A new antibiotic regimen treats and prevents intra-amniotic inflammation/infection in patients with preterm PROM. J Matern Fetal Neonatal Med. 2016 Sep;29(17):2727-37. doi: 10.3109/14767058.2015.1103729. Epub 2015 Dec 2. PMID 26441216
- [Result] Sgayer I, Francis YN, Miron D, Shprits E, Sheffer VF, Rechnitzer H, Lowenstein L, Wolf MF. Compared perinatal outcomes of two prophylactic antibiotic regimens for preterm premature rupture of membranes: a randomized controlled trial. Am J Obstet Gynecol MFM. 2023 May;5(5):100900. doi: 10.1016/j.ajogmf.2023.100900. Epub 2023 Feb 13. PMID 36791845